CLINICAL TRIAL: NCT06279091
Title: Correlation of Children and Parental Anxiety and Effectiveness of Breathing Exercises on Anxiety Reduction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Alaa Albakr, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A0104023PP
Record Dates: First submitted 2024-02-13; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Dental Anxiety
Keywords: Dental anxiety; Parental anxiety; Breathing Exercises; Bubble Blower Breathing; Diaphragmatic Breathing; Relaxation; Distruction

STUDY DESIGN:
Intervention Model Description: Selected children will be divided randomly into 3 groups:
  Control group (Group I). Diaphragmatic Breathing group (Group II). Bubble Blower Breathing group (Group III).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tell show do technique (Experimental): apply normal treatment with basic behavioral technique as a control group.
  Interventions: Behavioral: Tell Show Do
- Diaphragmatic breathing technique (Experimental): apply normal treatment with breathing exercises as relaxation and distruction technique to reduce the dental anxiety.
  Interventions: Behavioral: Diaphragmatic Breathing
- Bubble Blower breathing technique (Experimental): apply normal treatment with breathing exercises by bubbleblower which is a play therapy as relaxation and distruction technique to reduce the dental anxiety.
  Interventions: Behavioral: Bubble Blower Breathing

INTERVENTIONS:
Behavioral: Diaphragmatic Breathing — apply breathing exercises to evaluate the effectiveness on anxiety reduction
  Arms: Diaphragmatic breathing technique
Behavioral: Bubble Blower Breathing — apply breathing exercises by using bubble blower to evaluate the effectiveness on anxiety reduction
  Arms: Bubble Blower breathing technique
Behavioral: Tell Show Do — apply basic behavioral management technique as control group
  Arms: tell show do technique

SUMMARY:
The purpose of this study to evaluate the correlation between children and parental dental anxiety as well as to evaluate the effectiveness of breathing exercises on anxiety reduction.

DETAILED DESCRIPTION:
This study evaluated The Correlation of Children and Parental Anxiety and Effectiveness of Breathing Exercises on Anxiety Reduction

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5_8 years old.
* Moderate or severe dental anxiety based on the (CDAS).
* Good general health, free from any systemic diseases or psychological disorders.
* Teeth indicated for restoration treatment under local anesthesia.
* No allergy to anesthetic drugs

Exclusion Criteria:

* Use of analgesics before treatment.
* Presenting with acute pain and requiring emergency dental treatment.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2024-05-23 (Estimated)

PRIMARY OUTCOMES:
scale of dental anxiety by Corah Dental Anxiety Scale (CDAS) | up to 12 Weeks
  The CDAS is composed of four questions, with each question offering five possible responses. These responses are rated on a scale from 1 (representing no anxiety) to 5 (indicating extreme anxiety). The total anxiety score, which ranges from 4 to 20, is calculated by summing the scores from these questions. This scale categorizes anxiety levels as low (CDAS 4-8), moderate (CDAS 9-12), and high anxiety (CDAS 13-20).
  this scale used to evaluate correlation of children and parental anxiety.
scale of dental anxiety by Facial Image Scale (FIS) | up to 12 Weeks
  It consists of a single item with five response options, represented by faces ranging from severely happy(1) to very sad (5).
scale of dental anxiety by Venham Clinical Anxiety Scale (VCAS) | up to 12 Weeks
  This scale rates anxiety levels on a scale from 0 to 5. A score of 0 indicates relaxation, smiling, willingness, and the ability to converse. On the other hand, a score of 5 represents general loud crying and an inability to engage in verbal communication or cope with the situation.
scale of dental anxiety by Pulse Oximeter | up to 12 weeks
  To measure heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Albakr, Master, Principal Investigator — Researcher of Pediatric Dentistry Faculty of Dentistry Mansoura University; Salwa M Awad, Prof, Study Director — Prof. of Pediatric Dentistry and Dental Public Health Faculty of Dentistry Mansoura University; Rizk A Elagamy, PhD, Study Director — Assistant Professor of Pediatric Dentistry Faculty of Dentistry Mansoura University
Locations (1):
- Mansura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol to other Researchers
Supporting Information: Study Protocol
Time Frame: within 6 month
Access Criteria: for any one